CLINICAL TRIAL: NCT00210834
Title: A Randomized, Open-Label Study Of Epoetin Alfa (PROCRIT) Initiated At 40,000 Units Every Week Versus 80,000 Units Every Two Weeks In Anemic Patients With Cancer Receiving Chemotherapy
Brief Title: An Efficacy and Safety Study of Epoetin Alfa (PROCRIT) Initiated at 40,000 Units Every Week Versus 80,000 Units Every Two Weeks in Anemic Patients With Cancer Receiving Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004633
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-05

CONDITIONS: Anemia
Keywords: PROCRIT, Erythropoietin, Epoetin alfa, Hemoglobin level
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The primary objective of this study is to compare end of study hemoglobin levels between Epoetin alfa at 40,000 units administered subcutaneously once every week and at 80,000 units subcutaneously every two weeks in anemic patients with cancer receiving chemotherapy. The secondary objectives of the study are to assess the Hb response, time to Hb response, transfusion requirements, and safety.

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center study to compare end of study hemoglobin level between Epoetin alfa (PROCRIT) at 40,000 units administered subcutaneously once every week (qw) and at 80,000 units subcutaneously every two weeks (q2w) in approximately 280 anemic patients with cancer receiving chemotherapy. The study hypothesis is that a dosing regimen of PROCRIT 80,000 Units q2w subcutaneously (sc) is non-inferior to a dosing regimen of PROCRIT 40,000 Units qw sc with respect to the change in hemoglobin (Hb) from baseline to Study Week 13 for patients with chemotherapy associated anemia and this respective dosing regimen is generally well-tolerated. The patients will receive subcutaneous (under the skin) injections of Epoetin alfa (PROCRIT) at one of the following dosing regimens: 1- Starting dose of 40,000 units sc qw (once every week) OR 2- Starting dose of 80,000 units sc q2w (every two weeks)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-myeloid malignancy
* Baseline hemoglobin value of <= 11 g/dL unrelated to transfusion
* Planned chemotherapy for a minimum of 12 weeks during the study
* Life expectancy of >= 6 months
* ECOG Performance Status 0-2

Exclusion Criteria:

* Diagnosis of a myeloid malignancy or known history of myelodysplasia
* Planned non-palliative radiation during the study
* Anemia due to factors other than cancer/chemotherapy
* Prior treatment with Epoetin alfa or any other erythropoietic agent within the previous three months
* History of uncontrolled cardiac arrhythmias or history of pulmonary emboli, deep vein thrombosis, ischemic stroke, other arterial or venous thrombotic events (excluding superficial thromboses), or known history of chronic coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2004-05; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The end of study Hb. The end of study Hb is defined as the patient's final Hb level, taken 2 weeks after the last dose of PROCRIT or at Week 13, whichever comes first.

SECONDARY OUTCOMES:
Time to 1 g/dL HB increase; Proportion of patients achieving a >= 1 g/dL Hb increase by week for Weeks 5-13; Time to Hb increase of 2 g/dL or achieving Hb of >= 12 g/dL; Proportion of patients achieving a >= 2 g/dL Hb increase or Hb of 12 g/dL by EOS

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Henry DH, Gordan LN, Charu V, Wilhelm FE, Williams D, Xie J, Woodman RC. Randomized, open-label comparison of epoetin alfa extended dosing (80 000 U Q2W) vs weekly dosing (40 000 U QW) in patients with chemotherapy-induced anemia. Curr Med Res Opin. 2006 Jul;22(7):1403-13. doi: 10.1185/030079906X115559. PMID 16834839
- See also: A Randomized, Open-Label Study of PROCRIT (Epoetin alfa) Initiated at 40,000 Units Every Week Versus 80,000 Units Every Two Weeks in Anemic Patients with Cancer Receiving Chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=612&filename=CR004633_CSR.pdf